CLINICAL TRIAL: NCT04138771
Title: Validation of an Artificial Intelligence System for Postoperative Management of Cataract Patients: A Clinical Trial
Brief Title: Validation of an Artificial Intelligence System for Postoperative Management of Cataract Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government); Xidian University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCPMOH2019-China-5
Record Dates: First submitted 2019-10-23; First posted 2019-10-24 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Cataract; Postoperative Complications; Artificial Intelligence
Keywords: Conjunctival hyperemia; Pterygium; Intraocular lens dislocation; Posterior capsule opacification; Pupil malformation; Suppurative endophthalmitis
MeSH Terms: conditions — Cataract; Postoperative Complications; Pterygium; Pupil Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients for AI test (Experimental): Device: an artificial intelligence system for postoperative management of cataract patients. These patients are enrolled in primary healthcare units and the AI clinic at Zhongshan Ophthalmic Center.
  Interventions: Device: An artificial intelligence system for postoperative management of cataract patients

INTERVENTIONS:
Device: An artificial intelligence system for postoperative management of cataract patients — This system can detect multiple postoperative complications of cataract patients and then provide a management strategy.

SUMMARY:
Cataract surgery is the current standard of management for cataract patients, which is typically succeeded by a postoperative follow-up schedule. Here, the investigators established and validated an artificial intelligence system to achieve automatic management of postoperative patients based on analyses of visual acuity, intraocular pressure and slit-lamp images. The management strategy can also change according to postoperative time.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had surgery of cataract extraction combined with introcular lens implantation.
* Patients should be aware of the contents and signed for the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01-01; Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of accurate, mistaken and miss detection of this artificial intelligence diagnostic system. | Up to 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China